CLINICAL TRIAL: NCT00296621
Title: Efficacy Study of Oral Glutamine Supplementation in Duchenne Muscular Dystrophy
Brief Title: Effect of Oral Glutamine on Muscle Mass and Function in Duchenne Muscular Dystrophy
Acronym: MDB-GLN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Régis Hankard, MD PhD, CHU de Poitiers
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: P030420; AOM 03 121
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: glutamine; nutrition; children; pediatrics; randomized controlled clinical trial; therapy; supplement; oral administration; handicap
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: L-Glutamine
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: L-Glutamine — L-Glutamine
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether long-term oral glutamine supplementation is effective in improving muscle mass and function in children with Duchenne muscular dystrophy (DMD).

DETAILED DESCRIPTION:
Glutamine inhibits whole body protein degradation in children with Duchenne Muscular Dystrophy (DMD). The effect is observed after 5 h oral glutamine administration and is also found when glutamine is given over a 10-day period. This multi-site national study aims to evaluate the functional benefit of long-term oral glutamine administration in 30 DMD children using a randomized double-blind placebo-controlled cross-over design. The study includes two 4-month periods: 1) a treatment period in which the subject receives oral glutamine (0.5 g/kg/d) and 2) a control period in which the subject receives a placebo. The order of treatment allocation is randomized. The two 4-month periods are separated by a 1 month wash-out period. The children are monitored every 2 months during period 1 (M0, M2, M4) and period 2 (M5, M7, M9) in the clinical investigation centres of Hospital Robert Debré in Paris and the CHR&U de Lille, as well as the clinical research centre of the CHU de Poitiers. Evidence of a functional benefit would involve evaluating the administration of glutamine over longer periods (as early as possible following diagnosis) among severely handicapped children and in other chronic pathologies associated with increased muscle protein catabolism. In DMD, such evidence would enable children to undergo gene therapy under improved physical condition.

Comparisons: Glutamine administration compared to placebo on the following outcome measures: walking speed on a standard course, work (kcal) and power (kcal/s) in relation to effort, body composition (bioelectrical impedance analysis and BIPHOTONIC absorptiometry), muscle mass (24-h urinary creatinine excretion), indices of protein degradation (CPK and 3-methyl histidine excretion) and biochemical parameters (electrolytes, fasting glucose, transaminases, insulin, IgfI, Igf-BPI).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Duchenne muscular dystrophy
* Able to walk >170 m
* Absence of hepatic insufficiency
* Absence of renal insufficiency

Exclusion Criteria:

* Dependent upon wheelchair
* Body weight >60kg
* Liver failure
* Kidney failure
* Surgery scheduled during the year following the first visit

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-02; Primary Completion 2008-02 (Estimated); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
walking speed at 0,2,4,5,7,9 months | at 0,2,4,5,7,9 months

SECONDARY OUTCOMES:
work (kcal) at 0,2,4,5,7,9 months | at 0,2,4,5,7,9 months
power (kcal/s) at 0,2,4,5,7,9 months | at 0,2,4,5,7,9 months
2-minute walk test at 0,2,4,5,7,9 months | at 0,2,4,5,7,9 months
body composition (bioelectrical impedance analysis) at 0,2,4,5,7,9 months | at 0,2,4,5,7,9 months
body composition (BIPHOTONIC absorptiometry) at 4,9 months | at 4,9 months
muscle mass (24-h urinary creatinine excretion) at 0,2,4,5,7,9 months | at 0,2,4,5,7,9 months
indices of protein degradation (CPK and 3-methyl histidine excretion) at 0,2,4,5,7,9 months | at 0,2,4,5,7,9 months
biochemical parameters (electrolytes, fasting glucose, transaminases, insulin, IgfI, Igf-BP3) at 0,2,4,5,7,9 months | at 0,2,4,5,7,9 months

CONTACTS AND LOCATIONS:
Overall Officials: Régis Hankard, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire (CHU) de Poitiers
Locations (5):
- France (5):
  - Centre d'Investigation Clinique, Hôpital Cardiologique, CHR&U de Lille, Lille
  - Service d'Hépato Gastro Entérologie, Hôpital Jeanne de Flandre, CHR&U de Lille, Lille
  - Service de Neuropédiatrie, Hôpital Roger Salengro, CHR&U de Lille, Lille
  - Centre d'Investigation Clinique (CIC9202), Hôpital Robert Debré, Assistance Publique-Hôpitaux de Paris, Paris
  - Pédiatrie Multidisciplinaire et Nutrition de l'Enfant, Centre Hospitalier Universitaire de Poitiers, Poitiers

REFERENCES:
- [Background] Mok E, Eleouet-Da Violante C, Daubrosse C, Gottrand F, Rigal O, Fontan JE, Cuisset JM, Guilhot J, Hankard R. Oral glutamine and amino acid supplementation inhibit whole-body protein degradation in children with Duchenne muscular dystrophy. Am J Clin Nutr. 2006 Apr;83(4):823-8. doi: 10.1093/ajcn/83.4.823. PMID 16600934
- [Background] Hankard R, Mauras N, Hammond D, Haymond M, Darmaun D. Is glutamine a 'conditionally essential' amino acid in Duchenne muscular dystrophy? Clin Nutr. 1999 Dec;18(6):365-9. doi: 10.1016/s0261-5614(99)80017-x. PMID 10634922
- [Background] Hankard RG, Hammond D, Haymond MW, Darmaun D. Oral glutamine slows down whole body protein breakdown in Duchenne muscular dystrophy. Pediatr Res. 1998 Feb;43(2):222-6. doi: 10.1203/00006450-199802000-00011. PMID 9475288
- [Background] Hankard RG, Haymond MW, Darmaun D. Effect of glutamine on leucine metabolism in humans. Am J Physiol. 1996 Oct;271(4 Pt 1):E748-54. doi: 10.1152/ajpendo.1996.271.4.E748. PMID 8897864
- [Background] Hankard RG, Darmaun D, Sager BK, D'Amore D, Parsons WR, Haymond M. Response of glutamine metabolism to exogenous glutamine in humans. Am J Physiol. 1995 Oct;269(4 Pt 1):E663-70. doi: 10.1152/ajpendo.1995.269.4.E663. PMID 7485479
- [Background] Mok E, Beghin L, Gachon P, Daubrosse C, Fontan JE, Cuisset JM, Gottrand F, Hankard R. Estimating body composition in children with Duchenne muscular dystrophy: comparison of bioelectrical impedance analysis and skinfold-thickness measurement. Am J Clin Nutr. 2006 Jan;83(1):65-9. doi: 10.1093/ajcn/83.1.65. PMID 16400051
- [Derived] Mok E, Letellier G, Cuisset JM, Denjean A, Gottrand F, Alberti C, Hankard R. Lack of functional benefit with glutamine versus placebo in Duchenne muscular dystrophy: a randomized crossover trial. PLoS One. 2009;4(5):e5448. doi: 10.1371/journal.pone.0005448. Epub 2009 May 6. PMID 19421321